CLINICAL TRIAL: NCT01782235
Title: A Randomized, Double-blind, Parallel, Placebo-controlled Trial to Evaluate the Efficacy of Tocilizumab for the Treatment of Primary Sjögren's Syndrome.
Brief Title: Efficacy of Tocilizumab in Primary Sjögren's Syndrome.
Acronym: ETAP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5206; 2012-002045-37 (EudraCT Number)
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Primary Sjögren's Syndrome (pSS)
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Tocilizumab arm (Experimental): Tocilizumab arm will receive tocilizumab.
  Interventions: Drug: Tocilizumab
- Placebo arm (Placebo Comparator): Placebo arm will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab
  Arms: Tocilizumab arm
Drug: Placebo
  Arms: Placebo arm

SUMMARY:
Primary Sjögren's syndrome (pSS) is a systemic autoimmune disease characterized by lymphocytic infiltration leading to destruction of acinar and ductal cells and loss of glandular parenchyma. The main symptoms of pSS are dry eyes and dry mouth, diffuse pain, and fatigue. One third of patients develop systemic features, the most severe being lymphomas.

Serum IL-6 is increased in serum, saliva, and tears of patients with pSS. IL-6 plays a pivotal role in B-cell activation, a hallmark of the pathogenesis of pSS, and in T-cell differentiation. Tocilizumab, a recombinant humanised monoclonal antibody acts as an IL-6R antagonist. The aim of this randomised double blind placebo controlled trial iss to evaluate the efficacy of tocilizumab for the treatment of pSS.

ELIGIBILITY:
Inclusion Criteria :

* Patient with primary Sjögren's syndrome according to the European - American consensus group criteria.
* ESSDAI score ≥ 5.
* In women in childbearing age, effective contraception during treatment and 3 months following treatment discontinuation.

Exclusion Criteria:

* Patient with previous history of therapy with tocilizumab.
* Prednisone treatment introduced two weeks before inclusion or a change in this drug dose within two weeks before inclusion.
* A prednisone dose ≥ 15 mg per day.
* Non-steroidal anti-inflammatory drugs, pilocarpine hydrochloride, cyclosporine, cimeviline if introduced within two weeks before inclusion.
* Therapy with methotrexate, Hydroxychloroquine, chloroquine, quinacrine, leflunomide, psychoactive drug if introduced within 8 weeks before inclusion or a dose change within 8 weeks before inclusion.
* Treatment with azathioprine or mycophenolate mofetil within 8 weeks before inclusion.
* Live and live attenuated vaccines given within 4 weeks before inclusion.
* Any biologic treatment within 6 month before inclusion.
* Treatment with cyclophosphamide, intravenous immunoglobulin therapy or plasmapharese therapy in the last 6 months before inclusion.
* Systemic auto-immune disease.
* Patient with previous history of diverticular perforations, complications of diverticulitis, peritonite or inflammatory bowel disease (such as Crohn's disease and Colitis ulcerative).
* Patient with history of severe infection within 4 weeks before inclusion.
* Patient with history of infection within 2 weeks before inclusion.
* Patient with chronic infection or infection returns (e.g. tuberculose, VHB, VHC…).
* Positive serology tests for HIV, HBV, HCV.
* Severe uncontrolled dyslipidemia.
* Hepatocellular insufficiency.
* Unstable cardiovascular disease.
* Severe or chronic kidney disease, severe or chronic lung disease, severe or chronic endocrine disorder, severe or chronic neurological disease ( not related to the SJP).
* Patient with history of solid organ transplantation or haematopoietic stem cell transplantation.
* Patient with history of lymphoma, neoplasia diagnosed 5 years before inclusion except squamous and basal cell cancers and carcinoma in situ of the uterine cervix.
* Severe complications of SJp at the inclusion: vasculitis with renal neurologic, digestive or cardiac involvement, interstitial lung disease, symptomatic cryoglobulinemia with severe neurologic involvement, renal function impairment, severe myositis, corticotherapy ≥ 1 mg/kg in the last 30 days before inclusion.
* Neutropenia < 1000*10^6 .
* Thrombocytopenia < 50 000/µl
* ALT or AST > 3 x ULN
* alcohol and drug addiction : withdrawal at least one year before inclusion
* A major surgical procedure in the 8 weeks before inclusion or a scheduled major surgery
* Pregnant woman, breast feeding woman
* Adults under supervision or guardianship
* Patient taking part in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-07-24 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Improvement of the ESSDAI score equal to or greater than 3 points compared to enrollment. | 24 weeks
  Improvement of the ESSDAI score equal to or greater than 3 points compared to enrollment, with no new domain with high activity of the ESSDAI compared to enrollment, and no clinical worsening according to the clinician (no worsening compared to enrollment greater than 1 point of the Systemic Activity 0-10 VAS according to the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques-Eric Gottenberg, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

REFERENCES:
- [Result] Felten R, Devauchelle-Pensec V, Seror R, Duffau P, Saadoun D, Hachulla E, Pierre Yves H, Salliot C, Perdriger A, Morel J, Mekinian A, Vittecoq O, Berthelot JM, Dernis E, Le Guern V, Dieude P, Larroche C, Richez C, Martin T, Zarnitsky C, Blaison G, Kieffer P, Maurier F, Dellal A, Rist S, Andres E, Contis A, Chatelus E, Sordet C, Sibilia J, Arnold C, Tawk MY, Aberkane O, Holterbach L, Cacoub P, Saraux A, Mariette X, Meyer N, Gottenberg JE. Interleukin 6 receptor inhibition in primary Sjogren syndrome: a multicentre double-blind randomised placebo-controlled trial. Ann Rheum Dis. 2021 Mar;80(3):329-338. doi: 10.1136/annrheumdis-2020-218467. Epub 2020 Nov 18. PMID 33208345